CLINICAL TRIAL: NCT06890715
Title: A Randomized, Open-label, Two-period, Double-crossover Comparative Pharmacokinetic (PK) Study of a Single Oral Dose of Ramelteon Modified-Release Tablets and Ramelteon Tablets in Chinese Healthy Subjects
Brief Title: Comparative Pharmacokinetic Study of Ramelteon Modified-Release Tablets and Ramelteon Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Beijing CTSmed Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CTS-CO-2545
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Insomnia Characterized
Keywords: Ramelteon; Modified-Release; Chronic insomnia characterized by difficulties in falling asleep or maintaining sleep; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group T (Experimental): Test product (T): Ramelteon Modified-Release Tablets Strength: 8 mg/tablet Batch No.: G12308010 Content: 8 mg/tablet Valid to: 2025-8-16 Storage Conditions:Not higher than 25°C, sealed store Manufacturer: Overseas Pharmaceuticals, Ltd.
  Interventions: Drug: Test product (T): Ramelteon Modified-Release Tablets
- Group R (Active Comparator): Reference product (R): Ramelteon Tablets Strength: 8 mg/tablet Batch No.: 12216533 Content: 8 mg/tablet Valid to: 2024-10 Storage Conditions: 25 ° C (77°F) storage, allowing short-term temperature deviations of 15-30 ° C (59-86°F) Manufacturer:Takeda Pharmaceuticals America, Inc.
  Interventions: Drug: Reference product (R): Ramelteon Tablets

INTERVENTIONS:
Drug: Test product (T): Ramelteon Modified-Release Tablets — Oral, take 1 tablet at a time, once a day.
  Arms: Group T
Drug: Reference product (R): Ramelteon Tablets — Oral, take 1 tablet at a time, once a day.
  Arms: Group R

SUMMARY:
A randomized, open-label, two-period, double-crossover comparative pharmacokinetic (PK) study of a single oral dose of Ramelteon Modified-Release Tablets and Ramelteon Tablets in Chinese healthy subjects Primary objective: To evaluate the bioequivalence of the test product and the reference product by comparing their plasma concentrations and main PK parameters by oral administration in healthy Chinese subjects using Ramelteon Modified-Release Tablets (strength: 8 mg/tablet) developed by Overseas Pharmaceuticals, Ltd. as the test product and Ramelteon Tablets (trade name: Rozerem®, strength: 8 mg/tablet) produced by Takeda Pharmaceuticals America, Inc. as the reference product. Secondary objective: To evaluate the safety of Ramelteon Modified-Release Tablets (test product) and Ramelteon Tablets (reference product) with oral administration after drinking milk in healthy Chinese subjects.

DETAILED DESCRIPTION:
The trial was divided into screening period, period I, period II and safety follow-up period. The washout period is 2 days during the period.

Screening period: All subjects must sign an informed consent prior to participating in the trial. Screening tests were performed from Day -14 to Day 1 of administration.

Period I: 12 qualified subjects were screened and admitted to the Phase I ward of the Clinical Research Center on Day-1. After being reviewed and confirmed by the investigators, they were randomly divided into 2 groups, T-R group and R-T group, with 6 participants in each group. The normal diet was set at 8:00, 12:00 and 18:00 on the day of administration, and the uniform diet was required during the trial. After dinner at 18:00, all subjects were given 120mL whole milk starting at 21:57, one test product (Ramelteon Modified-Release Tablets (strength: 8 mg/tablet) or one reference product (Ramelteon Tablets (trade name: Rozerem®, strength: 8 mg/tablet) , and 120mL of warm water, the subject can lie down half after taking the drug, had no water within 1 hour after taking the drug, and fasted until breakfast the next day. PK blood samples were collected according to the time required by the scheme.

Period II : With a washout period of 2 days, the subjects underwent the period II of administration and blood collection on the night of Day 3, and the trial method in period II is the same as that in period I.

Vital signs (including body temperature, respiration, pulse, and blood pressure) were measured 1 hour before administration, at 2.0±0.5h, 5.0±0.5h, and 24.0±1.0h after each period of administration. Subjects were hospitalized throughout the trial period and underwent physical examination, vital signs measurement, electrocardiogram, and laboratory-related tests on Day 3 after the period II of dosing (female subjects were required to undergo blood pregnancy tests). Subject Lelt the stage I ward after completing PK sampling and the above examination.

Safety Follow-up: During the Day 8-Day 11 period, subjects will be contacted by telephone to collect information on drug combinations and adverse events after discharge from the study center.

Blood sample collection and processing: Cubital venous blood will be collected at 29 time points: before administration (0 h) (within 1.0h before administration) and 20min, 40min, 1h, 1h20min, 1h40min, 2h, 2h20min, 2h40min, 3h, 3h20min, 3h40min, 4h, 4h20min, 4h40min, 5h, 5h20min, 5h40min, 6h, 6h20min, 6h40min, 7h, 7h20min, 7h40min, 8h, 9h, 10h, 12h and 24h after administration of each period, and 4.0mL of blood was drawn and placed in the labeled EDTA-2K anticoagulant vacuum blood collection tube. Immediately after blood collection, the sampling vessels were gently and completely reversed three times and mixed with anticoagulant and temporarily placed at room temperature until centrifugation, centrifuged at 4℃ (set at 2-8 ℃) at 1700g for 10min. After centrifugation, the samples were removed from the centrifuge, and the plasma was collected and divided into two tubes (detection tube and backup tube) with corresponding labels. The test tube is about 0.8mL, and the remaining plasma is loaded into the backup tube. Blood samples were collected from the beginning, centrifugation was completed within 60 minutes, and plasma was frozen at -20 ° C (-30 ° C ~-10 ° C) or -80 ° C (-90 ° C ~-60 ° C) within 120 minutes. Samples stored in the -20 ° C refrigerator were transferred to the -80 ° C refrigerator for storage after 24 hours of blood collection. After the collection of blood samples of all subjects, the plasma samples of the detection tube will be transferred to the analysis and testing center for blood concentration determination, and the plasma samples of the backup tube will be stored in the clinical research unit or a third party designated by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 45 years (including 18 and 45 years);
2. Male subjects with a body weight ≥ 50.0 kg, and female subjects with a body weight ≥ 45.0 kg; BMI (BMI = body weight (kg)/[height (m)]2) within the range of 19-26.0 kg/m2 (including the critical value);
3. Subject who fully understands the purpose, nature, method and possible adverse reactions of the study, voluntarily acts as a subject, and signs informed consent prior to the commencement of any study procedure;;
4. Subjects who are able to communicate well with the investigator and understand and adhere to the study requirements.

Exclusion Criteria:

1. Subjects with an allergic history to the study drug or other melatonin or any other component of the study drug, or an allergic history to drug, food , pollen or a specific allergic history (asthma, allergic rhinitis);
2. Subjects who have special dietary requirements and cannot accept a unified diet;
3. Subjects with a history of dysphagia or any gastrointestinal disorder affecting drug absorption;
4. Subjects who cannot tolerate venipuncture , or with needle fainting or blood collection difficulties;
5. Subjects with clinically significant hematological, endocrine, cardiovascular, hepatic, renal and pulmonary disorders that may affect drug absorption, distribution, metabolism and excretion;
6. Vital signs examination, physical examination, clinical laboratory examination (blood routine, urine routine, blood biochemistry, coagulation four, pregnancy test (female), etc.), 12-lead electrocardiogram, chest X-ray examination results judged by researchers to be clinically significant;
7. Subjects with a surgical history within the 3 months prior to the study or taking the study drug or who plan to have surgery during the trial ；
8. Those who received the vaccine within 28 days before the first dose； 9) Subjects with blood donation or massive blood loss (> 450 mL) within 3 months before the study;

10) Subjects taking special diet (including pitaya or grapefruit and products containing grapefruit ingredients) or having strenuous exercise within 7 days before taking the study drug, or having other factors affecting drug absorption, distribution, metabolism and excretion; 11) Subjects administered with any prescription drugs, over-the-counter, herbal, or health products within 14 days prior to taking the study drug; 12) Drug users with a history of interaction with rametylamine tablets within 30 days prior to screening (fluvoxamine, rifampicin, ketoconazole, fluconazole, Donepezil, doxepin, Zolpidem, etc.; 13) Regular drinkers within 6 months prior to the study, i.e., drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirit containing 40% alcohol or 150 mL of wine); 14) Subjects who have a history of smoking in the first 3 months of prior to screening; Or who cannot stop using any tobacco products during the test period; Or positive results of tobacco test; 15) Subjects who have consumed chocolate, any caffeine-containing, or xanthine-rich food or beverage, such as coffee, strong tea, and cola 48 h before taking the study drug; 16) Subjects having taken any alcohol-containing products within 48 h before taking the study drug, or having a positive result for alcohol screening; Subjects positive for drug screening or with a history of drug abuse within the past five years or using drugs 3 months before the trial; 17) Female subjects with positive pregnancy test or lactating during the screening period or during the trial;Subjects (including male subjects) had a birth plan or could not use effective contraception from 2 weeks before the trial screening to 1 month after the trial ended; 18) Subjects positive for HBsAg, HCV-Ab, anti-HIV or primary syphilis screening; 19) Subjects who have participated in other clinical trials and used experimental drugs or devices within 3 months prior to screening; 20) Subjects with underlying medical, psychiatric, psychological or other discomfort conditions, poor compliance, or who, as judged by the investigator, are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual ramelteon and ramelteon metabolite M-II plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual ramelteon and ramelteon metabolite M-II plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual ramelteon and ramelteon metabolite M-II plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai He Associate Chief Pharmacist, Doctor, Principal Investigator — The Zhujiang Hospital of Southern Medical University
Locations (1):
- clinical trial centre of Medical ethics committee of Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No